CLINICAL TRIAL: NCT02870322
Title: Measuring the Feasibility of Fruit and Vegetable or Recreation Prescriptions Among UW-Madison Students
Brief Title: Fruit And Vegetable Or Recreation Prescriptions for UW-Madison Students
Acronym: FAVORx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0372; 1K24AT006543-01 (NIH)
Record Dates: First submitted 2016-07-28; First posted 2016-08-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; lifestyle prescription; prevention; physical activity; healthy eating
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fruit and Vegetable CSA Prescription (Active Comparator): Study participants randomized to the "CSA group" will be expected to pick up their weekly CSA box at University Health Services and to commit to using and consuming as much of the produce as they are able. CSA group participants will also be required to attend two cooking and food preparation classes coordinated by Slow Food UW. The classes will teach study participants how to properly clean and prepare the fruits and vegetables from a weekly CSA box, and also offer techniques and show them how to cook the foods in a healthy manner. These classes will also educate study participants on the benefits of eating fruits and vegetables and buying them from local farmers. These two classes will only exist for study participants in this fruit and veggie CSA group. Participants in the "CSA group" will also be required to take a field trip to the farm providing their CSA share, which will offer the opportunity for participants to gain a better understanding of from where their food comes.
  Interventions: Behavioral: Fruit and Vegetable CSA Prescription
- Bikeshare Prescription (Active Comparator): Study participants randomized to the "bikeshare group" will be expected to use B-cycle bikes for transportation and/or recreation as much as is safe and appropriate. Bikeshare group participants will be required to attend one bicycle use/safety course. This course will introduce the B-cycle program, demonstrate use of the B-cycle station, provide information use of helmets and safety gear, and provide information on the basics of cycling and keeping yourself safe and comfortable while riding in traffic. The study participants in this group will also be required to attend a class on the benefits of exercise, including bicycling, among other forms of physical activity. This class will be offered by the University Health Services Wellness program. B-cycle usage, including estimated distance traveled and frequency of use, will be tracked via the B-cycle Madison website.
  Interventions: Behavioral: Bikeshare Prescription
- Control (No Intervention): Study participants in the control group will receive continued "usual care" from University Health Services providers, which includes educational brochures on healthy eating and exercising, plus a cash payment. Control group participants are not part of a wait-list group.

INTERVENTIONS:
Behavioral: Fruit and Vegetable CSA Prescription — Study Participants will collect and use fruit and vegetable CSA boxes given to them weekly for 10 weeks.
  Arms: Fruit and Vegetable CSA Prescription
Behavioral: Bikeshare Prescription — Study participants will use bikeshare for transportation and physical activity for 10 weeks
  Arms: Bikeshare Prescription

SUMMARY:
This research will use randomized controlled trial (RCT) methodology to assess the feasibility of a prescription for fruit/vegetable CSA shares or exercise by bikeshare on obesity-related outcomes. Three cohorts of n=10 University of Wisconsin-Madison (UW) students (total 30) will be randomized to three groups: (1) a 10-week fruit and vegetable community supported agriculture (CSA) share prescription program with vegetable education and cooking support from UW Slow Food; (2) a 10-week Madison B-cycle bikeshare membership prescription program with exercise support or (3) a non-interventional wait-list control group. The primary outcome will be change in Body Mass Index (BMI) (a measure of obesity using a person's weight in kilograms divided by his or her height in meters squared). Secondary outcomes will be fasting lipids, blood pressure, and glycated hemoglobin (HGA1c) levels. All of these measures will be tested at baseline and just after the 10-week intervention

DETAILED DESCRIPTION:
This research will use randomized controlled trial (RCT) methodology to assess the feasibility of a prescription by University Health Services (UHS) Providers for fruit/vegetable CSA shares or exercise by bikeshare on obesity-related outcomes. Three cohorts of n=10 UW-Madison students (total 30) will be randomized to three groups: (1) a 10-week fruit and vegetable community supported agriculture (CSA) share prescription program with vegetable education and cooking support from UW Slow Food; (2) a 10-week Madison B-cycle bikeshare membership prescription program with exercise support from the UHS wellness program; or (3) a non-interventional wait-list control group. The primary outcome will be change in Body Mass Index (a measure of obesity using a person's weight in kilograms divided by his or her height in meters squared). Secondary outcomes will be fasting lipids, blood pressure, and HGA1c levels. All of these measures will be tested at baseline and just after the 10-week intervention. Fasting lipids and HGA1c levels will be assessed through a blood draw. Study participants will be asked to refrain from eating or drinking anything except for water 8-12 hours prior to the blood draw. Study participants will fill out validated questionnaires assessing perceived stress, physical activity levels, self-efficacy, social support, and general mental and physical health at baseline and after the intervention. Study participants will also conduct a 3 day dietary recall before and after the intervention.

Study participants randomized to the "CSA group" will be expected to pick up their weekly CSA box at University Health Services and to commit to using and consuming as much of the produce as they are able. CSA group participants will also be required to attend two cooking and food preparation classes coordinated by Slow Food UW. The classes will teach study participants how to properly clean and prepare the fruits and vegetables from a weekly CSA box, and also offer techniques and show them how to cook the foods in a healthy manner. These classes will also educate study participants on the benefits of eating fruits and vegetables and buying them from local farmers. These two classes will only exist for study participants in this fruit and veggie CSA group. Participants in the "CSA group" will also be required to take a field trip to the farm providing their CSA share, which will offer the opportunity for participants to gain a better understanding of from where their food comes.

Study participants randomized to the "bikeshare group" will be expected to use B-cycle bikeshare bicycles for transportation and/or recreation as much as is safe and appropriate. Bikeshare group participants will be required to attend two bicycle use/safety courses. These courses will introduce the B-cycle program, demonstrate use of the B-cycle station, provide information use of helmets and safety gear, and provide information on the basics of cycling and keeping yourself safe and comfortable while riding a B-cycle bike in traffic. B-cycle usage, including estimated distance traveled and frequency of use, will be tracked via the B-cycle Madison website.

Study participants in the control group will receive continued "usual care" from University Health Services providers, which includes educational brochures on healthy eating and exercising. Control group participants are not part of a wait-list group.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 years of age or older
2. Seeking healthcare from UW UHS
3. Is enrolled at UW-Madison for next academic year
4. BMI >25
5. Living off-campus for following year, and not with parents or guardians
6. Basic English fluency and literacy

Exclusion Criteria:

1. Currently exercises more than 2 times per week for 30 minutes or more
2. Participant is pregnant or plans to be pregnant
3. Regularly rides a bicycle (more than 1-2 times per month)
4. Currently participates or has already participated in a fruit /vegetable CSA share

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Between Baseline and Follow-Up visits for a total of 16-18 weeks
  Change in Body Mass Index in kg/m^2 will be calculated using the participant weight (kg) and height (meters) measured at Baseline and Follow-Up visits, which will be approximately a 16-18 week timeframe over the intervention period.

SECONDARY OUTCOMES:
Fasting Lipid Panel | Baseline, 12 - 16 weeks
  Fasting Lipid Panel will be collected at Baseline and at Follow-Up, which will be approximately a 12-16 week timeframe.
Glycated Hemoglobin (HgA1c) | Baseline, 12 -16 weeks
  Glycated Hemoglobin will be collected at Baseline and at Follow-Up, which will be approximately a 12-16 week timeframe.
Blood Pressure | Baseline, 12 - 16 weeks
  Blood Pressure will be taken at Baseline and at Follow-Up, which will be approximately a 12-16 week timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce P Barrett, MD, PhD, Principal Investigator — Professor, Clinician
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No